CLINICAL TRIAL: NCT00614614
Title: Immunogenicity and Safety Study of a Booster Dose of GSK Biologicals' Meningococcal Vaccine 134612 Given at 12-15 Months of Age or at 15-18 Months of Age (Co-administered With Infanrix®) in Primed Healthy Toddlers.
Brief Title: Immuno,Safety of GSK Vaccine 134612 Given at Age of 12-15 Months 15-18 Months Post-priming With GSK Vaccine 792014
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 110870; 110871 (Other: GSK)
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2012-07-20 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2016-10

CONDITIONS: Infections, Meningococcal
Keywords: Meningococcal disease; Toddlers; Neisseria meningitidis; Meningococcal vaccines; Immunogenicity; Human serum bactericidal assay; Safety; Vaccines, conjugate; Booster vaccination
MeSH Terms: conditions — Meningococcal Infections | interventions — Hib-MenCY-TT vaccine; Diphtheria-Tetanus-acellular Pertussis Vaccines; Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate; PEDIARIX

STUDY DESIGN:
Who Masked: Care Provider

ARMS (2):
- Menhibrix 1 Group (Experimental): Subjects received 3 doses of Menhibrix vaccine and 3 doses of Pediarix vaccine at 2, 4 and 6 months of age during the Primary Vaccination Phase. For the Booster Vaccination Phase, subjects were re-randomized and received either 1 dose of Nimenrix vaccine (at 12-15 months of age) and 1 dose of Infanrix vaccine (at 15-18 months of age) [Nimenrix 1 Group] or a fourth dose of Menhibrix vaccine (at 12-15 months of age) and 1 dose of Infanrix vaccine (at 15-18 months of age) [Menhibrix 2 Group], or 1 dose of Nimenrix vaccine co-administered with 1 dose of Infanrix vaccine (at 15-18 months of age) [Nimenrix 2 Group].
  Interventions: Biological: GSK Biologicals' Meningococcal vaccine GSK134612 (Nimenrix); Biological: GSK Biologicals' Hib-meningococcal vaccine GSK 792014 (Menhibrix); Biological: Infanrix®; Biological: Pediarix®
- ActHIB- Infanrix Group (Active Comparator): Subjects received 3 doses of ActHIB vaccine and 3 doses of Pediarix vaccine at 2, 4 and 6 months of age and 1 booster dose of Infanrix vaccine at 15-18 months of age.
  Interventions: Biological: Infanrix®; Biological: ActHIB®; Biological: Pediarix®

INTERVENTIONS:
Biological: GSK Biologicals' Meningococcal vaccine GSK134612 (Nimenrix) — One dose in the booster phase as intramuscular injection
  Other Names: Nimenrix
  Arms: Menhibrix 1 Group
Biological: GSK Biologicals' Hib-meningococcal vaccine GSK 792014 (Menhibrix) — Three doses in the priming phase and, for Menhibrix 2 Group, one dose in the booster phase as intramuscular injection
  Other Names: Menhibrix
  Arms: Menhibrix 1 Group
Biological: Infanrix® — One dose as intramuscular injection
Biological: ActHIB® — Three doses in the priming phase as intramuscular injection
  Arms: ActHIB- Infanrix Group
Biological: Pediarix® — Three doses in the priming phase as intramuscular injection

SUMMARY:
The purpose of the study is to characterize the immunogenicity & safety of a booster dose of GSK Biologicals' meningococcal vaccine 134612 given at 12-15 months of age or at 15-18 months of age (co-administered with Infanrix®) in healthy toddlers primed with GSK Biological's Hib-meningococcal vaccine 792014. This study is single-blinded for the primary phase and open-label for the booster phase.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the titer of antibody for serogroups A, C, Y and W-135 and the safety of a booster dose of GSK Biologicals' meningococcal vaccine 134612 given to toddlers who were primed with GSK Biological's Hib-meningococcal vaccine 792014. In addition, this study will provide immunogenicity and safety data on the co-administration of Infanrix with meningococcal vaccine 134612 as compared to Infanrix administered alone.

Depending on the group the subject is assigned to, one or two blood samples will be taken out of the subject's arm during the study.

The protocol posting has been updated following a protocol amendment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects for whom the investigator believes that parents/guardians can and will comply with the requirements of the protocol.
* A male or female between, and including, 6 and 12 weeks of age (+ 6 days) at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born after 36 weeks gestation.
* For inclusion in the booster phase, subjects must have received all three doses in the primary phase.

Exclusion Criteria:

Exclusion criteria for enrolment (primary phase)

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of study vaccine(s).
* Previous vaccination against Neisseria meningitidis, Haemophilus influenzae type b, diphtheria, tetanus, pertussis, and/or poliovirus; more than one previous dose of hepatitis B vaccine.
* History of Neisseria meningitidis, hepatitis B, Haemophilus influenzae type b, diphtheria, tetanus, polio or pertussis diseases.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, or by dry natural latex rubber.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at time of enrollment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Concurrent participation in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).

Exclusion criteria for enrolment (booster phase)

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding entry into the booster phase (Visit 4), or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days of entry into the booster phase (Visit 4) with the exception of Prevnar® and Hib (see the following three criteria) (Note; licensed influenza vaccine is allowed throughout the study)
* Planned administration/administration of a fourth dose of Prevnar® within 30 days of a booster dose of Infanrix®
* Previous administration of a booster dose of Hib prior to entry to the booster phase.
* Previous administration of a primary dose of Hib vaccine that is not part of the study protocol.
* Previous vaccination against Neisseria meningitidis that is not part of the study protocol.
* Previous vaccination with diphtheria, tetanus and pertussis antigens outside of the primary phase of the study.
* History of Neisseria meningitidis, Hib, diphtheria, tetanus or pertussis diseases.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, or by dry natural latex rubber.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at time of enrollment.
* Administration of immunoglobulins and/or any blood products within the past 3 months or planned administration during the study period.
* Concurrent participation in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1558 (Actual)
Dates: Start 2008-02-13; Primary Completion 2009-07-31 (Actual); Study Completion 2009-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (53):
- United States (53):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Benton, Arkansas
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, West Des Moines, Iowa
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Bossier City, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Niles, Michigan
  - GSK Investigational Site, Portage, Michigan
  - GSK Investigational Site, Richland, Michigan
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Clyde, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Huber Heights, Ohio
  - GSK Investigational Site, Gresham, Oregon
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Greenville, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Provo, Utah
  - GSK Investigational Site, Roy, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, St. George, Utah
  - GSK Investigational Site, Syracuse, Utah
  - GSK Investigational Site, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Leonardi M, Latiolais T, Sarpong K, Simon M, Twiggs J, Lei P, Rinderknecht S, Blatter M, Bianco V, Baine Y, Friedland LR, Baccarini C, Miller JM. Immunogenicity and reactogenicity of Infanrix when co-administered with meningococcal MenACWY-TT conjugate vaccine in toddlers primed with MenHibrix and Pediarix. Vaccine. 2015 Feb 11;33(7):924-32. doi: 10.1016/j.vaccine.2014.09.064. Epub 2014 Oct 8. PMID 25305567
- [Derived] Leonardi M, Latiolais T, Sarpong K, Simon M, Twiggs J, Lei P, Rinderknecht S, Blatter M, Bianco V, Baine Y, Friedland LR, Miller JM. Quadrivalent meningococcal (MenACWY-TT) conjugate vaccine or a fourth dose of H. influenzae-N. meningitidis C/Y conjugate vaccine (HibMenCY-TT) is immunogenic in toddlers who previously received three doses of HibMenCY-TT in infancy. Vaccine. 2015 Feb 11;33(7):933-41. doi: 10.1016/j.vaccine.2014.08.027. Epub 2014 Aug 21. PMID 25152325
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 110870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1558 subjects (1276 in the Menhibrix 1 Group and 282 in ActHIB- Infanrix Group) were enrolled; however, 4 of these subjects never received vaccine. Thus, 1554 subjects (1272 in the Menhibrix 1 Group and 282 in ActHIB- Infanrix Group) were vaccinated during primary vaccination phase.
Groups:
- ActHIB- Infanrix Group: Subjects received 3 doses of ActHIB vaccine and 3 doses of Pediarix vaccine at 2, 4 and 6 months of age at Primary Vaccination Phase and 1 booster dose of Infanrix vaccine at 15-18 months of age at Booster Vaccination Phase.
- Nimenrix 1 Group: Subjects received 1 dose of Nimenrix vaccine at 12-15 months of age and 1 dose of Infanrix vaccine at 15-18 months of age during Booster Vaccination Phase.
- Menhibrix 2 Group: Subjects received a fourth dose of Menhibrix vaccine at 12-15 months of age and 1 dose of Infanrix vaccine at 15-18 months of age during Booster Vaccination Phase.
- Nimenrix 2 Group: Subjects received 1 dose of Nimenrix vaccine co-administered with 1 dose of Infanrix vaccine at 15-18 months of age during Booster Vaccination Phase.
Period: Primary Vaccination Phase
Arm/Group | Menhibrix 1 Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Started | 1272 | 282 | 0 (Primary vaccination phase involved subjects from MenHibrix 1 Group and ActHIB- Infanrix Group only.) | 0 (Primary vaccination phase involved subjects from MenHibrix 1 Group and ActHIB- Infanrix Group only.) | 0 (Primary vaccination phase involved subjects from MenHibrix 1 Group and ActHIB- Infanrix Group only.)
Completed | 1182 | 265 | 0 (Primary vaccination phase involved subjects from MenHibrix 1 Group and ActHIB- Infanrix Group only.) | 0 (Primary vaccination phase involved subjects from MenHibrix 1 Group and ActHIB- Infanrix Group only.) | 0 (Primary vaccination phase involved subjects from MenHibrix 1 Group and ActHIB- Infanrix Group only.)
Not Completed | 90 | 17 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 45 | 6 | 0 | 0 | 0
Not completed — Lost to Follow-up | 26 | 8 | 0 | 0 | 0
Not completed — Protocol Violation | 9 | 3 | 0 | 0 | 0
Not completed — Other | 4 | 0 | 0 | 0 | 0
Period: Booster Vaccination Phase
Arm/Group | Menhibrix 1 Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Started | 0 (Menhibrix 1 Group was re-randomized to Nimenrix 1,Menhibrix 2 and Nimenrix 2 Groups in booster phase) | 233 | 432 | 229 | 409
Completed | 0 (Menhibrix 1 Group was re-randomized to Nimenrix 1,Menhibrix 2 and Nimenrix 2 Groups in booster phase) | 227 | 405 | 210 | 396
Not Completed | 0 | 6 | 27 | 19 | 13
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 3 | 4
Not completed — Lost to Follow-up | 0 | 5 | 17 | 10 | 8
Not completed — Protocol Violation | 0 | 0 | 2 | 3 | 0
Not completed — Other | 0 | 1 | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Menhibrix 1 Group: Subjects received 3 doses of Menhibrix vaccine and 3 doses of Pediarix vaccine at 2, 4 and 6 months of age during Primary Vaccination Phase.
- Total: Total of all reporting groups
Arm/Group | Menhibrix 1 Group | ActHIB- Infanrix Group | Total
Number analyzed (Participants) | 1272 | 282 | 1554
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.6 (1.25) | 8.7 (1.25) | 8.6 (1.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 606 | 150 | 756
  Male | 666 | 132 | 798
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage / African American | 135 | 20 | 155
  American Indian or Alaskan native | 4 | 0 | 4
  Asian - Central/South Asian heritage | 4 | 0 | 4
  Asian - East Asian heritage | 4 | 1 | 5
  Asian - Japanese heritage | 1 | 1 | 2
  Asian - South East Asian heritage | 8 | 2 | 10
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  White - Arabic / North African heritage | 14 | 3 | 17
  White - Caucasian / European heritage | 974 | 223 | 1197
  Unspecified | 127 | 32 | 159

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serum Bactericidal Activity Using Human Complement (hSBA) Antibody Titers for N. Meningitidis Serogroups A(MenA), W-135(MenW-135), C(MenC) and Y(MenY) Greater Than or Equal to Protocol Specified Cut-off Value in Nimenrix 1 Group
Description: The cut-off values assessed for hSBA-MenA, hSBA-MenW-135, hSBA-MenC and hSBA-MenY were greater than or equal to (≥) 1:8
Time Frame: One month post vaccination at 12-15 months of age (Month 11)
Population: Analysis was performed on Booster According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available against at least one study vaccine antigen component during booster phase vaccination. Analysis was only performed on the Nimenrix 1 Group.
Measure: Count of Participants; unit: Participants
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 0 | 291 | 0 | 0
Participants
  hSBA-MenA: number analyzed (Participants) | 0 | 257 | 0 | 0
  hSBA-MenA |  | 254 |  |
  hSBA-MenC: number analyzed (Participants) | 0 | 286 | 0 | 0
  hSBA-MenC |  | 286 |  |
  hSBA-MenW-135: number analyzed (Participants) | 0 | 273 | 0 | 0
  hSBA-MenW-135 |  | 270 |  |
  hSBA-MenY |  | 291 |  |

2. Primary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenW-135, hSBA-MenC and hSBA-MenY Antibody Titers Greater Than or Equal to Protocol Specified Cut-off Value in Nimenrix 2 Group
Description: The cut-off values assessed for hSBA-MenA, hSBA-MenW-135, hSBA-MenC and hSBA-MenY were greater than or equal to (≥) 1:8
Time Frame: One month post vaccination at 15-18 months of age (Month 14)
Population: Analysis was performed on Booster According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available against at least one study vaccine antigen component during booster phase vaccination. Analysis was only performed on the Nimenrix 2 Group.
Measure: Count of Participants; unit: Participants
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 0 | 0 | 0 | 303
Participants
  hSBA-MenA: number analyzed (Participants) | 0 | 0 | 0 | 258
  hSBA-MenA |  |  |  | 248
  hSBA-MenC: number analyzed (Participants) | 0 | 0 | 0 | 293
  hSBA-MenC |  |  |  | 293
  hSBA-MenW-135: number analyzed (Participants) | 0 | 0 | 0 | 283
  hSBA-MenW-135 |  |  |  | 279
  hSBA-MenY |  |  |  | 303

3. Primary Outcome: Geometric Mean Antibody Titers for hSBA-MenC and hSBA-MenY in Nimenrix 1 Group
Description: Antibody titers were expressed as Geometric mean titers (GMTs)
Time Frame: One month post vaccination at 12-15 months of age (Month 11)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 0 | 291 | 0 | 0
titer
  hSBA-MenC: number analyzed (Participants) | 0 | 286 | 0 | 0
  hSBA-MenC |  | 3845.0 [3310.8 to 4465.4] |  |
  hSBA-MenY |  | 4800.9 [4162.0 to 5537.9] |  |

4. Primary Outcome: Geometric Mean Antibody Titers for hSBA-MenC and hSBA-MenY in Nimenrix 2 Group
Description: Antibody titers were expressed as Geometric mean titers (GMTs)
Time Frame: One month post vaccination at 15-18 months of age (Month 14)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 0 | 0 | 0 | 303
titer
  hSBA-MenC: number analyzed (Participants) | 0 | 0 | 0 | 293
  hSBA-MenC |  |  |  | 7230.5 [6244.1 to 8372.8]
  hSBA-MenY |  |  |  | 7487.6 [6604.4 to 8488.9]

5. Primary Outcome: Number of Subjects With Anti-Diptheria (Anti-D) and Anti-Tetanus (Anti-T) Antibody Concentrations Greater Than or Equal to Protocol Specified Cut-off Value in Nimenrix 2 Group and ActHIB- Infanrix Group
Description: The cut-off value assessed for Anti-D and Anti-T were greater than or equal to (≥) 1.0 International Units per milliliter (IU/mL).
Time Frame: One month post vaccination at 15-18 months of age (Month 14)
Population: Analysis was performed on Booster According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available against at least one study vaccine antigen component during booster phase vaccination. It was performed on the Nimenrix 2 and ActHIB- Infanrix Group.
Measure: Count of Participants; unit: Participants
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 146 | 0 | 0 | 254
Participants
  Anti-D | 146 |  |  | 253
  Anti-T: number analyzed (Participants) | 146 | 0 | 0 | 253
  Anti-T | 145 |  |  | 253

6. Primary Outcome: Geometric Mean Antibody Titers for hSBA-MenC and hSBA-MenY in Menhibrix 2 Group
Description: Antibody titers were expressed as Geometric mean titers (GMTs)
Time Frame: One month post vaccination at 12-15 months of age (Month 11)
Population: Analysis was performed on Booster According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available against at least one study vaccine antigen component during booster phase vaccination. Analysis was only performed on the Menhibrix 2 Group.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 0 | 0 | 157 | 0
titer
  hSBA-MenC: number analyzed (Participants) | 0 | 0 | 155 | 0
  hSBA-MenC |  |  | 2676.1 [2131.8 to 3359.5] |
  hSBA-MenY |  |  | 2227.7 [1881.9 to 2637.0] |

7. Primary Outcome: Number of Subjects With hSBA-MenC and hSBA-MenY Antibody Titers Greater Than or Equal to Protocol Specified Cut-off Value in Menhibrix 2 Group
Description: The cut-off values assessed for hSBA-MenC and hSBA-MenY were greater than or equal to (≥) 1:8
Time Frame: One month post vaccination at 12-15 months of age (Month 11)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 0 | 0 | 157 | 0
Participants
  hSBA-MenC: number analyzed (Participants) | 0 | 0 | 155 | 0
  hSBA-MenC |  |  | 155 |
  hSBA-MenY |  |  | 157 |

8. Primary Outcome: Geometric Mean Antibody Concentrations for Anti-PT (Pertusis Toxoid), Anti-FHA (Filamentous Hemagglutinin) and Anti-PRN (Pertactin) in Nimenrix 2 Group and ActHIB- Infanrix Group
Description: Concentrations were provided as Geometric mean concentrations (GMCs) and expressed as enzyme-linked immunosorbent assay units per milliliter (EL.U/mL)
Time Frame: One month after vaccination at 15-18 months of age (Month 14)
Population: Analysis was performed on Booster According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available against at least one study vaccine antigen component during booster phase vaccination. Analysis was performed on Nimenrix 2 and ActHIB- Infanrix Group.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 146 | 0 | 0 | 254
EL.U/mL
  Anti-PT | 91.0 [81.7 to 101.4] |  |  | 67.7 [62.0 to 73.9]
  Anti-FHA: number analyzed (Participants) | 146 | 0 | 0 | 253
  Anti-FHA | 422.9 [369.0 to 484.6] |  |  | 353.2 [320.8 to 388.9]
  Anti-PRN: number analyzed (Participants) | 146 | 0 | 0 | 253
  Anti-PRN | 315.1 [274.2 to 362.1] |  |  | 189.2 [167.2 to 214.1]

9. Secondary Outcome: Number of Subjects With hSBA-MenC and hSBA-MenY Antibody Titers Greater Than or Equal to Protocol Specified Cut-off Values in Nimenrix 1 Group and Menhibrix 2 Group
Description: The cut-off values assessed for hSBA-MenC and hSBA-MenY were greater than or equal to (≥) 1:4
Time Frame: One month after vaccination at 12-15 months of age (Month 11)
Population: Analysis was performed on Booster According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available against at least one study vaccine antigen component during booster phase vaccination. Analysis was performed on the Nimenrix 1 and Menhibrix 2 Group.
Measure: Count of Participants; unit: Participants
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 0 | 291 | 157 | 0
Participants
  hSBA-MenC: number analyzed (Participants) | 0 | 286 | 155 | 0
  hSBA-MenC |  | 286 | 155 |
  hSBA-MenY |  | 291 | 157 |

10. Secondary Outcome: Number of Subjects With hSBA-MenA and hSBA MenW-135 Antibody Titers Greater Than or Equal to Protocol Specified Cut-off Values in Nimenrix 1 Group
Description: The cut-off values assessed for hSBA-MenA and hSBA-MenW-135 were greater than or equal to (≥) 1:4
Time Frame: One month after vaccination at 12-15 months of age (Month 11)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 0 | 273 | 0 | 0
Participants
  hSBA-MenA: number analyzed (Participants) | 0 | 257 | 0 | 0
  hSBA-MenA |  | 256 |  |
  hSBA-MenW-135 |  | 270 |  |

11. Secondary Outcome: Geometric Mean Antibody Titers for hSBA-MenA and hSBA MenW-135 in Nimenrix 1 Group
Description: Antibody titers were expressed as Geometric mean titers (GMTs)
Time Frame: One month after vaccination at 12-15 months of age (Month 11)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 0 | 273 | 0 | 0
titer
  hSBA-MenA: number analyzed (Participants) | 0 | 257 | 0 | 0
  hSBA-MenA |  | 94.8 [84.1 to 106.9] |  |
  hSBA-MenW-135 |  | 923.9 [776.0 to 1099.9] |  |

12. Secondary Outcome: Geometric Mean Antibody Titers for hSBA-MenC and hSBA-MenY in Nimenrix 2 Group
Description: Antibody titers were expressed as Geometric mean titers (GMTs)
Time Frame: Prior to vaccination at 15-18 months of age (Month 13)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 0 | 0 | 0 | 268
titer
  hSBA-Men C |  |  |  | 67.6 [55.5 to 82.3]
  hSBA-MenY |  |  |  | 142.3 [121.1 to 167.2]

13. Secondary Outcome: Number of Subjects With hSBA-MenC and hSBA-MenY Antibody Titers Greater Than or Equal to Protocol Specified Cut-off Values in Nimenrix 2 Group
Description: The cut-off values assessed for hSBA-MenC and hSBA-MenY were greater than or equal to (≥) 1:4 and ≥ 1:8
Time Frame: Prior to vaccination at 15-18 months of age (Month 13)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 0 | 0 | 0 | 268
Participants
  hSBA-MenC ≥ 1:4 |  |  |  | 243
  hSBA-MenC ≥ 1:8 |  |  |  | 241
  hSBA-MenY ≥ 1:4 |  |  |  | 258
  hSBA-MenY ≥ 1:8 |  |  |  | 258

14. Secondary Outcome: Anti-D and Anti-T Geometric Mean Antibody Concentrations
Description: Concentrations were provided as Geometric Mean Concentrations(GMCs) and expressed as International Units per milliliter (IU/mL).
Time Frame: One month after vaccination with Infanrix at 15-18 months of age (Month 14)
Population: Analysis was performed on Booster According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available against at least one study vaccine antigen component during booster phase vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 146 | 252 | 132 | 254
IU/mL
  Anti-D | 8.259 [7.347 to 9.285] | 7.214 [6.592 to 7.895] | 7.360 [6.508 to 8.323] | 7.458 [6.820 to 8.155]
  Anti-T: number analyzed (Participants) | 146 | 252 | 132 | 253
  Anti-T | 5.500 [4.877 to 6.204] | 7.400 [6.900 to 7.936] | 8.458 [7.762 to 9.215] | 11.751 [10.818 to 12.765]

15. Secondary Outcome: Number of Subjects With Anti-D and Anti-T Antibody Concentrations Greater Than or Equal to Protocol Specified Cut-off Value
Description: The cut-off value assessed for Anti-D and Anti-T were greater than or equal to (≥) 0.1 International Units per milliliter (IU/mL).
Time Frame: One month after vaccination with Infanrix at 15-18 months of age (Month 14)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 146 | 252 | 132 | 254
Participants
  Anti-D | 146 | 252 | 132 | 254
  Anti-T: number analyzed (Participants) | 146 | 252 | 132 | 253
  Anti-T | 146 | 252 | 132 | 253

16. Secondary Outcome: Number of Subjects With Anti-PT, Anti-FHA and Anti-PRN Concentrations Greater Than or Equal to Protocol Specified Cut-off Value
Description: The cut-off values assessed were greater than or equal to (≥) 5 enzyme-linked immunosorbent assay units per milliliter (EL.U/mL)
Time Frame: One month after vaccination with Infanrix at 15-18 months of age (Month 14)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 146 | 252 | 132 | 254
Participants
  Anti-PT: number analyzed (Participants) | 146 | 252 | 130 | 254
  Anti-PT | 146 | 252 | 130 | 254
  Anti-FHA: number analyzed (Participants) | 146 | 252 | 132 | 253
  Anti-FHA | 146 | 252 | 132 | 253
  Anti-PRN: number analyzed (Participants) | 146 | 252 | 132 | 253
  Anti-PRN | 146 | 251 | 132 | 253

17. Secondary Outcome: Geometric Mean Antibody Concentrations for Anti-PT, Anti-FHA and Anti-PRN in Nimenrix 1 Group and Menhibrix 2 Group
Description: as for outcome 8
Time Frame: One month after vaccination at 15-18 months of age (Month 14)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 0 | 252 | 132 | 0
EL.U/mL
  Anti-PT: number analyzed (Participants) | 0 | 252 | 130 | 0
  Anti-PT |  | 73.3 [66.7 to 80.5] | 86.9 [75.7 to 99.8] |
  Anti-FHA |  | 321.6 [289.9 to 356.7] | 371.7 [321.5 to 429.7] |
  Anti-PRN |  | 203.8 [178.7 to 232.5] | 220.2 [183.7 to 264.0] |

18. Secondary Outcome: Number of Subjects With Anti-D and Anti-T Antibody Concentrations Greater Than or Equal to Protocol Specified Cut-off Value in Nimenrix 1 Group and Menhibrix 2 Group
Description: The cut-off values assessed for Anti-D and Anti-T were greater than or equal to (≥) 1.0 International Units per milliliter (IU/mL).
Time Frame: One month after vaccination at 15-18 months of age (Month 14)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 0 | 252 | 132 | 0
Participants
  Anti-D |  | 250 | 132 |
  Anti-T |  | 250 | 132 |

19. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibody Titers Greater Than or Equal to Protocol Specified Cut-off Values in Nimenrix 2 Group
Description: The cut-off values assessed for hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY were greater than or equal to (≥) 1:4
Time Frame: One month after vaccination at 15-18 months of age (Month 14)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 0 | 0 | 0 | 303
Participants
  hSBA-MenA: number analyzed (Participants) | 0 | 0 | 0 | 258
  hSBA-MenA |  |  |  | 253
  hSBA-MenC: number analyzed (Participants) | 0 | 0 | 0 | 293
  hSBA-MenC |  |  |  | 293
  hSBA-MenW-135: number analyzed (Participants) | 0 | 0 | 0 | 283
  hSBA-MenW-135 |  |  |  | 279
  hSBA-MenY |  |  |  | 303

20. Secondary Outcome: Geometric Mean Antibody Titers for hSBA-MenA and hSBA-MenW-135 in Nimenrix 2 Group
Description: Antibody titers were expressed as Geometric mean titers (GMTs)
Time Frame: One month after vaccination with Infanrix at 15-18 months of age (Month 14)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 0 | 0 | 0 | 283
titer
  hSBA-MenA: number analyzed (Participants) | 0 | 0 | 0 | 258
  hSBA-MenA |  |  |  | 92.4 [80.6 to 105.9]
  hSBA-MenW-135 |  |  |  | 1582.9 [1321.8 to 1895.5]

21. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Adverse Events (AEs) Following Each Dose With Nimenrix or Menhibrix Vaccine
Description: Any was defined as any solicited local symptom reported regardless of intensity grade. Grade 3 redness and swelling was greater than (>) 30 millimeter (mm) and grade 3 pain was subjects crying when limb was moved/spontaneously painful.
Time Frame: During the 8-day follow-up period (Day 0-7) after vaccination in the booster phase
Population: The analysis was performed on Booster Total Vaccinated cohort which included all subjects who had received a study vaccine during the booster phase and had symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 0 | 408 | 217 | 386
Participants
  Any pain |  | 156 | 104 | 170
  Grade 3 pain |  | 7 | 4 | 2
  Any redness |  | 171 | 90 | 169
  Grade 3 redness |  | 3 | 1 | 5
  Any swelling |  | 97 | 54 | 105
  Grade 3 swelling |  | 3 | 1 | 3

22. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General AEs in the Booster Phase
Description: Any fever was defined as axillary temperature greater than or equal to 38.0 degree centigrade i.e ≥38.0°C, grade 3 fever was axillary temperature > 40.0°C. For other symptoms, any was defined as occurrence of any general symptom regardless of intensity grade or relation to vaccination and grade 3 was defined as a general symptom that prevented normal activity. Related was a general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 8-day follow-up period (Day 0-7) after dose 4 and dose 5 vaccination
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 209 | 408 | 217 | 384
Participants
  Any drowsiness, Dose 4 | 79 | 171 | 97 | 161
  Grade3 drowsiness, Dose 4 | 1 | 7 | 6 | 8
  Related drowsiness, Dose 4 | 62 | 148 | 80 | 132
  Any fever, Dose4 | 14 | 46 | 23 | 37
  Grade3 fever, Dose 4 | 0 | 2 | 2 | 1
  Related fever, Dose 4 | 7 | 32 | 16 | 23
  Any irritability, Dose 4 | 114 | 230 | 128 | 218
  Grade3 irritability, Dose 4 | 7 | 13 | 11 | 12
  Related irritability, Dose4 | 90 | 202 | 106 | 188
  Any loss of appetite, Dose4 | 55 | 144 | 73 | 138
  Grade3 loss of appetite, Dose4 | 3 | 7 | 5 | 7
  Related loss of apetite, Dose4 | 42 | 115 | 55 | 105
  Any drowsiness, Dose 5: number analyzed (Participants) | 0 | 384 | 197 | 0
  Any drowsiness, Dose 5 |  | 132 | 67 |
  Grade3 drowsiness, Dose 5: number analyzed (Participants) | 0 | 384 | 197 | 0
  Grade3 drowsiness, Dose 5 |  | 7 | 6 |
  Related drowsiness, Dose 5: number analyzed (Participants) | 0 | 384 | 197 | 0
  Related drowsiness, Dose 5 |  | 114 | 60 |
  Any fever, Dose 5: number analyzed (Participants) | 0 | 384 | 197 | 0
  Any fever, Dose 5 |  | 34 | 16 |
  Grade 3 fever, Dose 5: number analyzed (Participants) | 0 | 384 | 197 | 0
  Grade 3 fever, Dose 5 |  | 0 | 0 |
  Related fever, Dose 5: number analyzed (Participants) | 0 | 384 | 197 | 0
  Related fever, Dose 5 |  | 23 | 12 |
  Any irritability, Dose 5: number analyzed (Participants) | 0 | 384 | 197 | 0
  Any irritability, Dose 5 |  | 195 | 103 |
  Grade 3 irritabiity, Dose 5: number analyzed (Participants) | 0 | 384 | 197 | 0
  Grade 3 irritabiity, Dose 5 |  | 12 | 8 |
  Related irritability, Dose 5: number analyzed (Participants) | 0 | 384 | 197 | 0
  Related irritability, Dose 5 |  | 171 | 99 |
  Any loss of appetite, Dose 5: number analyzed (Participants) | 0 | 384 | 197 | 0
  Any loss of appetite, Dose 5 |  | 117 | 62 |
  Grade 3 loss of appetite, Dose 5: number analyzed (Participants) | 0 | 384 | 197 | 0
  Grade 3 loss of appetite, Dose 5 |  | 2 | 5 |
  Related loss of appetite, Dose 5: number analyzed (Participants) | 0 | 384 | 197 | 0
  Related loss of appetite, Dose 5 |  | 86 | 53 |

23. Secondary Outcome: Number of Subjects Reporting Any Rash
Description: Examples of rash included hives, idiopathic thrombocytopenic purpura, petechiae.
Time Frame: From the first booster phase visit up to six months after the last vaccination (Month 10-13 up to Month 19-22)
Population: The analysis was performed on Booster Total Vaccinated cohort which included all subjects who had received a study vaccine during the booster phase.
Measure: Count of Participants; unit: Participants
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 233 | 432 | 229 | 409
Participants | 40 | 93 | 54 | 83

24. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Adverse Events (AEs) Following Vaccination With Infanrix Vaccine
Description: Any was defined as any solicited local symptom reported regardless of intensity grade. Grade 3 redness and swelling was > 30 millimeter (mm) and grade 3 pain was subjects crying when limb was moved/spontaneously painful.
Time Frame: During the 8-day follow-up period (Day 0-7) after vaccination in the booster phase
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 210 | 385 | 197 | 374
Participants
  Any pain | 99 | 145 | 99 | 156
  Grade 3 pain | 4 | 5 | 2 | 4
  Any redness | 121 | 175 | 102 | 171
  Grade 3 redness | 4 | 9 | 5 | 2
  Any swelling | 80 | 114 | 73 | 113
  Grade 3 swelling | 5 | 6 | 5 | 2

25. Secondary Outcome: Number of Subjects Reporting Any New Onset of Chronic Illness (NOCI) and Any Emergency Room (ER) Visits
Description: NOCIs include autoimmune disorders, asthma, type I diabetes and allergies. AEs prompting emergency room visits or physician visits are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: From the first booster phase visit up to six months after the last vaccination (Month 10-13 up to Month 19-22)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 233 | 432 | 229 | 409
Participants
  Any NOCI(s) | 13 | 19 | 11 | 18
  Any ER visit(s) | 29 | 73 | 49 | 76

26. Secondary Outcome: Number of Subjects Reporting Any New Onset of Chronic Illness (NOCI) and Any Emergency Room (ER) Visits
Description: as for outcome 25
Time Frame: From the first primary study dose up to/excluding the first booster study dose (Month 0 up to Month 10-13)
Population: The analysis was performed on Primary Total Vaccinated cohort which included all subjects who had received a study vaccine during the primary phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix 1 Group | ActHIB- Infanrix Group
Number analyzed (Participants) | 1272 | 282
Participants
  Any NOCI(s) | 128 | 29
  Any ER visit(s) | 293 | 55

27. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs) After the First or Single Booster Phase Vaccination
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: During a 31-day follow-up period (Day 0-30)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Groups:
- Menhibrix 2 Group: Subjects received a fourth dose of Menhibrix vaccine at 12-15 months of age and 1 dose of Infanrix vaccine at 15-18 months of age.during Booster Vaccination Phase.
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 233 | 432 | 229 | 409
Participants | 101 | 194 | 105 | 182

28. Secondary Outcome: Number of Subjects Reporting Any Unsolicited AEs in Nimenrix 1 Group and Menhibrix 2 Group After the Second Booster Phase Vaccination
Description: as for outcome 27
Time Frame: During the 31-day follow-up period (Day 0-30)
Population: The analysis was performed on Booster Total Vaccinated cohort which included all subjects who had received a study vaccine during the booster phase. Analysis was performed on the Nimenrix 1 and Menhibrix 2 Group.
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix 2 Group: Subjects received 1 dose of Nimenrix vaccine co-administered with 1 dose of Infanrix vaccine at 15-18 months of age.during Booster Vaccination Phase.
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 0 | 432 | 229 | 0
Participants |  | 167 | 79 |

29. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: From the first primary study dose up to/excluding the first booster study dose (Month 0 up to Month 10-13).
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix 1 Group | ActHIB- Infanrix Group
Number analyzed (Participants) | 1272 | 282
Participants
  Any SAE(s) | 58 | 14
  Related SAE(s) | 1 | 0

30. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: as for outcome 29
Time Frame: From the first booster phase visit up to six months after the last vaccination (Month 10-13 up to Month 19-22)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Number analyzed (Participants) | 233 | 432 | 229 | 409
Participants
  Any SAE(s) | 2 | 15 | 3 | 9
  Related SAE(s) | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed from Month 0 up to Month 19-22. Systematically and non-systematically assessed frequent adverse events were assessed during the 8 day (Day 0-7) and 31 day (Day 0-30) period respectively after booster vaccination.
Description: Participants at risk for systematically assessed adverse events (AEs) = Booster Total Vaccinated cohort with symptom sheet completed and for non-systematically assessed other (non-serious) AEs = Booster Total Vaccinated cohort. For serious AEs, participants at risk = Primary Total Vaccinated cohort and Booster Total Vaccinated cohort respectively.
  Other Adverse Events were not collected for Menhibrix 1 Group.
Arm/Group | Menhibrix 1 Group | ActHIB- Infanrix Group | Nimenrix 1 Group | Menhibrix 2 Group | Nimenrix 2 Group
Serious Adverse Events (participants affected / at risk) | 58/1272 | 14/282 | 15/432 | 3/229 | 9/409
Other Adverse Events (participants affected / at risk) | 0/0 | 181/233 | 387/432 | 211/229 | 337/409
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Menhibrix 1 Group (N=1272) | ActHIB- Infanrix Group (N=282) | Nimenrix 1 Group (N=432) | Menhibrix 2 Group (N=229) | Nimenrix 2 Group (N=409)
Bronchiolitis (Infections and infestations) | 9 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Dehydration (Metabolism and nutrition disorders) | 7 | 2 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Gastroenteritis (Infections and infestations) | 5 | 2 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Convulsion (Nervous system disorders) | 3 | 1 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Croup infectious (Infections and infestations) | 4 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Otitis media (Infections and infestations) | 1 | 3 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Pyrexia (General disorders) | 3 | 1 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 4 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Cellulitis (Infections and infestations) | 3 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Pneumonia (Infections and infestations) | 1 | 2 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Skull fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Apnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Otitis media acute (Infections and infestations) | 2 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Respiratory syncytial virus infection (Infections and infestations) | 2 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Subcutaneous abscess (Infections and infestations) | 2 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Sudden infant death syndrome (General disorders) | 2 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Viral infection (Infections and infestations) | 1 | 1 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Beta haemolytic streptococcal infection (Infections and infestations) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Bronchitis (Infections and infestations) | 0 | 1 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Cyanosis (Cardiac disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Febrile convulsion (Nervous system disorders) | 0 | 1 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Gastric volvulus (Gastrointestinal disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Hypotonia (Nervous system disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Influenza (Infections and infestations) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Irritability (General disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Meningitis viral (Infections and infestations) | 0 | 1 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Obstructive uropathy (Renal and urinary disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Pertussis (Infections and infestations) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Pyelonephritis (Infections and infestations) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Septic shock (Infections and infestations) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Tachycardia (Cardiac disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Urinary tract infection (Infections and infestations) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Urosepsis (Infections and infestations) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0/0 | 0/0 | 0/0 — SAE assessed from the first primary dose up to the end of the primary ESFU period (Month 0 upto Month 10-13) for MenHibrix 1 Group and ActHIB-Infanrix Group.
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0/233 | 1 | 0 | 1 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Abscess (Infections and infestations) | 0/0 | 0/233 | 1 | 0 | 0 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Acidosis (Metabolism and nutrition disorders) | 0/0 | 0/233 | 0 | 1 | 0 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Adenoidectomy (Surgical and medical procedures) | 0/0 | 0/233 | 1 | 0 | 0 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Encephalitis viral (Infections and infestations) | 0/0 | 0/233 | 0 | 1 | 0 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Floppy infant (Musculoskeletal and connective tissue disorders) | 0/0 | 0/233 | 0 | 0 | 1 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Gastroenteritis viral (Infections and infestations) | 0/0 | 0/233 | 0 | 0 | 1 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Herpes oesophagitis (Infections and infestations) | 0/0 | 1/233 | 0 | 0 | 0 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Pancytopenia (Blood and lymphatic system disorders) | 0/0 | 0/233 | 0 | 0 | 1 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 0/0 | 0/233 | 1 | 0 | 0 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Somnolence (Nervous system disorders) | 0/0 | 0/233 | 1 | 0 | 0 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0/233 | 0 | 0 | 1 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Thrombocytopenia (Blood and lymphatic system disorders) | 0/0 | 0/233 | 0 | 1 | 0 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Upper respiratory infection (Infections and infestations) | 0/0 | 0/233 | 0 | 1 | 0 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Wound infection (Infections and infestations) | 0/0 | 0/233 | 0 | 0 | 1 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Dehydration (Metabolism and nutrition disorders) | 0/0 | 0/233 | 5 | 0 | 2 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Otitis media (Infections and infestations) | 0/0 | 0/233 | 2 | 0 | 1 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Pneumonia (Infections and infestations) | 0/0 | 0/233 | 3 | 0 | 0 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/0 | 1/233 | 1 | 0 | 0 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0/233 | 1 | 1 | 0 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Febrile convulsion (Nervous system disorders) | 0/0 | 0/233 | 0 | 2 | 0 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Gastroenteritis (Infections and infestations) | 0/0 | 0/233 | 1 | 0 | 1 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Pyrexia (General disorders) | 0/0 | 0/233 | 1 | 0 | 1 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Respiratory syncitial virus bronchiolitis (Infections and infestations) | 0/0 | 0/233 | 1 | 0 | 1 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Staphylococcal infection (Infections and infestations) | 0/0 | 0/233 | 1 | 0 | 1 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Cellulitis (Infections and infestations) | 0/0 | 0/233 | 1 | 0 | 0 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Croup infectious (Infections and infestations) | 0/0 | 0/233 | 1 | 0 | 0 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
Viral infection (Infections and infestations) | 0/0 | 0/233 | 1 | 0 | 0 — SAE assessed from the first booster phase visit up to 6 months after the last booster phase vaccination (Month 10-13 up to Month 19-22).
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Menhibrix 1 Group (N=0) | ActHIB- Infanrix Group (N=233) | Nimenrix 1 Group (N=432) | Menhibrix 2 Group (N=229) | Nimenrix 2 Group (N=409)
Pain (General disorders) | 0 | 0/0 | 156/408 | 104/217 | 170/386 — Pain was experienced during the 8-day (Days0-7) post-vaccination period following each dose with Nimenrix or MenHibrix vaccine in the booster phase.
Redness (General disorders) | 0 | 0/0 | 171/408 | 90/217 | 169/386 — Redness was experienced during the 8-day (Days0-7) post-vaccination period following each dose with Nimenrix or MenHibrix vaccine in the booster phase.
Swelling (General disorders) | 0 | 0/0 | 97/408 | 54/217 | 105/386 — Swelling was experienced during the 8-day (Days0-7) post-vaccination period following each dose with Nimenrix or MenHibrix vaccine in the booster phase.
Pain (General disorders) | 0 | 99/210 | 145/385 | 99/197 | 156/374 — Pain was experienced during the 8-day (Days0-7) post-vaccination period with Infanrix vaccine in the booster phase.
Redness (General disorders) | 0 | 121/210 | 175/385 | 102/197 | 171/374 — Redness was experienced during the 8-day (Days0-7) post-vaccination period with Infanrix vaccine in the booster phase.
Swelling (General disorders) | 0 | 80/210 | 114/385 | 73/197 | 113/374 — Swelling was experienced during the 8-day (Days0-7) post-vaccination period with Infanrix vaccine in the booster phase.
Drowsiness (General disorders) | 0 | 79/209 | 171/408 | 97/217 | 161/384 — Symptom experienced at Dose 4 vaccination with Nimenrix [ for Nimenrix 1 Group], MenHibrix [ for MenHibrix 2 Group], Nimenrix co-administered with Infanrix [ for Nimenrix 2 Group] and Infanrix [ for ActHIB-Infanrix Group].
Fever (General disorders) | 0 | 14/209 | 46/408 | 23/217 | 37/384 — Symptom experienced at Dose 4 vaccination with Nimenrix [ for Nimenrix 1 Group], MenHibrix [ for MenHibrix 2 Group], Nimenrix co-administered with Infanrix [ for Nimenrix 2 Group] and Infanrix [ for ActHIB-Infanrix Group].
Irritability (General disorders) | 0 | 114/209 | 230/408 | 128/217 | 218/384 — Symptom experienced at Dose 4 vaccination with Nimenrix [ for Nimenrix 1 Group], MenHibrix [ for MenHibrix 2 Group], Nimenrix co-administered with Infanrix [ for Nimenrix 2 Group] and Infanrix [ for ActHIB-Infanrix Group].
Loss of appetite (General disorders) | 0 | 55/209 | 144/408 | 73/217 | 138/384 — Symptom experienced at Dose 4 vaccination with Nimenrix [ for Nimenrix 1 Group], MenHibrix [ for MenHibrix 2 Group], Nimenrix co-administered with Infanrix [ for Nimenrix 2 Group] and Infanrix [ for ActHIB-Infanrix Group].
Drowsiness (General disorders) | 0 | 0/0 | 132/384 | 67/197 | 0/0 — Symptom experienced at Dose 5 vaccination with Infanrix vaccine for Nimenrix 1 Group and MenHibrix 2 Group.
Fever (General disorders) | 0 | 0/0 | 34/384 | 16/197 | 0/0 — Symptom experienced at Dose 5 vaccination with Infanrix vaccine for Nimenrix 1 Group and MenHibrix 2 Group.
Irritability (General disorders) | 0 | 0/0 | 195/384 | 103/197 | 0/0 — Symptom experienced at Dose 5 vaccination with Infanrix vaccine for Nimenrix 1 Group and MenHibrix 2 Group.
Loss of appetite (General disorders) | 0 | 0/0 | 117/384 | 62/197 | 0/0 — Symptom experienced at Dose 5 vaccination with Infanrix vaccine for Nimenrix 1 Group and MenHibrix 2 Group.
Otitis media (Infections and infestations) | 0 | 9 | 54 | 24 | 21 — Symptom experienced during the 31-day (Days 0-30) period after the first or single booster phase vaccination in all groups corresponding to Booster phase of study.
Upper respiratory tract infection (Infections and infestations) | 0 | 11 | 34 | 22 | 36 — Symptom experienced during the 31-day (Days 0-30) period after the first or single booster phase vaccination in all groups corresponding to Booster phase of study.
Otitis media (Infections and infestations) | 0 | 0/0 | 27 | 13 | 0/0 — Symptom experienced during the 31-day (Days 0-30) period after the second booster phase vaccination in Nimenrix 1 Group and MenHibrix 2 Group.
Upper respiratory tract infection (Infections and infestations) | 0 | 0/0 | 27 | 13 | 0/0 — Symptom experienced during the 31-day (Days 0-30) period after the second booster phase vaccination in Nimenrix 1 Group and MenHibrix 2 Group.
Diarrhoea (Gastrointestinal disorders) | 0 | 0/0 | 13 | 13 | 0/0 — Symptom experienced during the 31-day (Days 0-30) period after the second booster phase vaccination in Nimenrix 1 Group and MenHibrix 2 Group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.